CLINICAL TRIAL: NCT03092609
Title: Neuroplasticity in an Extended Amygdala Network as a Target Mechanism for Attention Bias Modification Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Michigan University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS13-555; R15MH110951 (NIH)
Record Dates: First submitted 2017-03-14; First posted 2017-03-28 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Anxiety
Keywords: Attentional Bias to Threat
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Bias Modification (Experimental)
  Interventions: Behavioral: Attention Bias Modification
- Attention Control (Active Comparator)
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Attention Bias Modification — Attention bias modification (ABM) sessions will consist of a modified dot-probe task that only contains incongruent trials (i.e., target-dot - neutral stimulus 100% pairing).
  Arms: Attention Bias Modification
Behavioral: Attention Control — Attention control (AC) sessions, will consist of a standard dot-probe task (i.e., target-dot - neutral/threat stimulus 50% pairing). Thus, for AC participants, bias should remain the same, while ABM participants should show a reduced bias to threat.
  Arms: Attention Control

SUMMARY:
Anxiety disorders are one of the most common psychological disorders. Underlying anxiety is an increased attentional bias to threat, which has been identified as a causal contributor in the development of anxiety. Given this causal relationship, attention bias modification was introduced as a treatment option where anxiety is reduced by training individuals to direct their attention away from threat and thereby decreasing anxiety. Over a decade of research using this approach, called attention bias modification (ABM), suggests that overall the approach is effective in reducing anxiety. Although ABM appears to be a very promising treatment option for anxiety, there are several factors limiting the effectiveness of ABM. These include the recognition of individual-level needs and a known underlying mechanism of action by which ABM is effective. Neuroimaging evidence suggests that attentional bias to visual threat is associated with a network of brain regions including the amygdala, anterior cingulate cortex, and visual cortex. In human participants, experience-dependent neuroplasticity is visible in voxel-based morphometry based measures of gray matter volume following training. Recently, voxel-based morphometry measures of gray matter volume have been linked to dendritic spine density-a known cellular mechanism for learning-related neuroplasticity. Thus, voxel-based morphometry measures are ideally suited to measure learning-related neuroplasticity following attention bias modification. In this proposal participants' level of attentional bias, anxiety, and gray matter volume will be measured before and after completing six weeks of attention bias modification training (N = 50) or attention control training (N= 50). The proposal aims to (1) establish that pre-treatment bias predicts variability in gray matter volume in the extended amygdala and anterior cingulate cortex, (2) assess the extent to which reduced extended amygdala and anterior cingulate cortex gray matter volume following ABM underlies reductions in attentional bias and anxiety, and (3) Establish pre-treatment bias as a predictor of successful ABM as measured by reduced bias, reduced anxiety, and reduced gray matter volume in the extended amygdala and anterior cingulate cortex. Consistent with the objectives of the AREA grant and NIMH's focus on identifying and validating new targets for treatment development that underlie disease mechanisms, the current proposal plans to involve students at a rural primarily undergraduate university in a research project aimed at establishing neuroplasticity in the extended amygdala and anterior cingulate cortex as a target mechanism for ABM training outcome, which could be used to objectively track training-related outcomes in anxiety treatment.

ELIGIBILITY:
Inclusion Criteria:

* Handedness (right handed)
* Normal Vision
* High Anxiety
* Preexisting Attentional Bias

Exclusion Criteria:

* No MRI contraindications
* No History of Head Injury
* No Neurological History
* Psychological History
* Limited Recreational Drug Use, No Abuse
* Limited Prescription Drug Use, No Abuse
* No Claustrophobia
* Not Pregnant

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Attentional Bias | Baseline and after 6 weeks of the intervention
  Reaction time difference to congruent and incongruent trials in the dot-probe task, which measure heightened attentional bias to threat.

SECONDARY OUTCOMES:
State and Trait Anxiety | Baseline and after 6 weeks of the intervention
  Anxiety as measured by the Speilberger State-Trait Anxiety Inventory

OTHER OUTCOMES:
MRI measures of gray matter volume | Baseline and after 6 weeks of the intervention
  T1-weighted MRI measures of gray matter volume
MRI measures of structural and functional connectivity | Baseline and after 6 weeks of the intervention
  Diffusion-tensor weighted MRI based measures of structural connectivity and functional MRI based measures of functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Carlson, PhD, Principal Investigator — Northern Michigan University
Locations (1):
- Northern Michigan University, Marquette, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the NIMH Data Archive

REFERENCES:
- [Derived] Carlson JM, Fang L, Koster EHW, Andrzejewski JA, Gilbertson H, Elwell KA, Zuidema TR. Neuroplastic changes in anterior cingulate cortex gray matter volume and functional connectivity following attention bias modification in high trait anxious individuals. Biol Psychol. 2022 Jul;172:108353. doi: 10.1016/j.biopsycho.2022.108353. Epub 2022 May 13. PMID 35569575
- [Derived] Carlson JM, Fang L. Attentional bias to threat and gray matter volume morphology in high anxious individuals. Cogn Affect Behav Neurosci. 2022 Jun;22(3):600-609. doi: 10.3758/s13415-021-00968-9. Epub 2021 Nov 9. PMID 34755317